CLINICAL TRIAL: NCT04885725
Title: Association Between Knee Isokinetic Testing and Lower Limb Functional Performance and Limb Symmetry
Acronym: Pro-knee
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Principal Investigator, Physician in the Sport Medicine Department (MD), PhD student, University Hospital, Caen
Other Study IDs: Pro-knee
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Proprioceptive Disorders
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: All group — All the participants performed the isokinetic proprioception and strength tests and the functional tests, on the same visit.

SUMMARY:
This study aimed to evaluate the association between the isokinetic knee strength and/or proprioception performance with the functional performance on the functional Hop-tests and Y-balance test.

This study included 20 healthy individuals who performed an isokinetic assessment of knee proprioception (joint position sense, JPS and threshold to detection of passive motion, TDPM) and flexors/extensors strength. At the same time, they performed a functional testing consisting of three Hop-tests (single, triple and cross-over) and the Lower Quarter Y-Balance Test (YBT-LQ). We tested the correlation between the isokinetic and functional performances, and limb symmetry indexes.

ELIGIBILITY:
Inclusion Criteria:

* individuals under 45 years of age who performed at least 4 hours of physical activity per week.

Exclusion Criteria:

* individuals unable to perform isokinetic muscle tests
* individuals with a current or recent lower limb injury with time loss from sport participation within the previous month
* individuals with previous severe knee injury (eg. Severe ligament tear, knee fracture)
* individuals taking medications with potential balance/coordination side effects.

Age Groups: Child, Adult, Older Adult
Study Population: Young healthy adults who volunteered to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
Strength | one evaluation at a single point in time through study completion, an average of 4 months
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer.
Knee proprioception, JPS1 | one evaluation at a single point in time through study completion, an average of 4 months
  Measurement of knee proprioception by the passive repositioning technique (JPS, in degrees) on isokinetic dynamometer.
Knee proprioception, JPS2 | one evaluation at a single point in time through study completion, an average of 4 months
  Measurement of knee proprioception by the active repositioning technique (JPS, in degrees) on isokinetic dynamometer.
Knee proprioception, TDPM | one evaluation at a single point in time through study completion, an average of 4 months
  Measurement of knee proprioception by the Threshold to Detection of Passive Motion (TDPM in degrees) on isokinetic dynamometer.
Functional testing, Hop tests | one evaluation at a single point in time through study completion, an average of 4 months
  Hop test. Single hop: Patients are instructed to stand on one leg and perform 1 jump as far as possible, landing on the same leg.
  The total distance is recorded (in cm) .Triple hop: Patients are instructed to stand on one leg and perform 3 hops as far as possible, landing on the same leg.
  The total distance for 3 consecutive hops is recorded (in cm). Cross-over hop test : The patient hops forward 3 times while alternately crossing over a marking The patient is instructed to position themselves such that the first of the 3 hops was lateral with respect to the direction of crossover The total distance hopped forward is recorded (in cm)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France